CLINICAL TRIAL: NCT03193060
Title: A Multi-centre, Prospective, Observational Study on Effectiveness and Safety of ZOLADEX® (Goserelin Acetate Implant) 10.8 mg and ZOLADEX® (Goserelin Acetate Implant) 3.6 mg in Chinese Patients With Localized or Locally Advanced Hormonal Treatment -naïve Prostate Cancer
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D8664R00001
Record Dates: First submitted 2017-05-08; First posted 2017-06-20 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Localized or Locally Advanced Prostate Cancer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a multi-centre, prospective observational study. The study plans to enrol 500 patients with localized or locally advanced prostate cancer who are eligible and intended to be prescribed Zoladex® (goserelin acetate implant) 10.8 mg or Zoladex® (goserelin acetate implant) 3.6 mg as monotherapy or in combination with androgen blockade (CAB) at 50 clinical sites in China. The effectiveness and safety data will be collected at baseline and each visit within 26 weeks after treatment of Zoladex®.

DETAILED DESCRIPTION:
Androgen Deprivation Therapy (ADT) is a standard treatment for locally advanced or metastatic prostate cancer. It is also increasingly used in patients with high-risk localized prostate cancer or in patients with prostate-specific antigen (PSA) relapse after local therapy.

The luteinizing hormone-releasing hormone (LHRH) agonists, such as goserelin acetate(Zoladex®), have provided an effective and reversible means of suppressing androgen level. Zoladex® was originally formulated as a 3.6mg depot injection. Goserelin acetate 10.8-mg depot, given once every 3 months, is pharmacodynamically equivalent to 3 consecutive monthly injections of the goserelin acetate 3.6-mg depot, offers a more convenient and cost-effective dosing regimen for patients.

Goserelin acetate 10.8-mg depot has been available in China since 2012. However, data on the effectiveness and safety of the long-acting depot of Zoladex® (goserelin acetate depot) 10.8mg specifically in a Chinese population is limited. A "real-world" observational study is proposed to establish the effectiveness and safety profile of Zoladex ® 10.8mg in Chinese patients with localized or locally advanced prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide informed consent, complete all study assessments and have complete medical record;
2. Male aged 18 years and over;
3. Diagnosis of localized or locally advanced prostate cancer requiring immediate hormonal therapy;
4. Being prescribed Zoladex ® (goserelin acetate implant) 10.8 mg or Zoladex ® (goserelin acetate implant) 3.6 mg in accordance with the terms of marketing authorization as monotherapy or in combination with androgen blockade (CAB);
5. More than 26 weeks' life expectancy;

Exclusion Criteria:

1. Patients who are planned to receive radiation therapy;
2. Patients with hypersensitivity to LHRH, its analogues, or any components of goserelin depot;
3. Previous or concurrent hormonal therapy including surgical castration, androgen blockers, oestrogen therapy, or other LHRH agonists.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with localized or locally advanced prostate cancer who are prescribed Zoladex® (goserelin acetate implant) 10.8 mg or 3.6 mg as monotherapy or in combination with androgen blockade (CAB), either as first line treatment or adjuvant therapy to radical prostatectomy (RP) are eligible to be the study target population.
Sampling Method: Non-Probability Sample
Enrollment: 308 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2019-12-27 (Actual); Study Completion 2019-12-27 (Actual)

PRIMARY OUTCOMES:
PSA level | each visit within 26 weeks during treatment
  Change from baseline in PSA level at each visit within 26 weeks during treatment
Serum Testosterone | each visit within 26 weeks during treatment
  Change from baseline in the serum Testosterone at each visit within 26 weeks during treatment

SECONDARY OUTCOMES:
Mean serum Testosterone level | each visit within 26 weeks during treatment
  Mean serum Testosterone level at baseline and each visit within 26 weeks during treatment
Mean serum PSA level | each visit within 26 weeks during treatment
  Mean serum PSA level at baseline and each visit within 26 weeks during treatment
Number of patients with serum Testosterone less than 50 ng/ml | each visit within 26 weeks during treatment
  Number of patients with serum Testosterone less than 50 ng/ml at each visit within 26 weeks during treatment
Incidence of Adverse Events (AEs) | each visit within 26 weeks during treatment
  Incidence of Adverse Events (AEs)
Incidence of AESI (cardiovascular related AE, sexual related AE) | each visit within 26 weeks during treatment
  Incidence of AESI (cardiovascular related AE, sexual related AE)
Incidence of Adverse Drug Reactions (ADRs) | each visit within 26 weeks during treatment
  Incidence of Adverse Drug Reactions (ADRs)
Incidence of AEs leading to treatment discontinuation | each visit within 26 weeks during treatment
  Incidence of AEs leading to treatment discontinuation
Proportion of patients with serum Testosterone less than 50 ng/ml | each visit within 26 weeks during treatment
  Proportion of patients with serum Testosterone less than 50 ng/ml at each visit within 26 weeks during treatment
Incidence of Serious Adverse Events (SAEs) | each visit within 26 weeks during treatment
  Incidence of Serious Adverse Events (SAEs)

CONTACTS AND LOCATIONS:
Locations (18):
- China (18):
  - Research Site, Beijing
  - Research Site, Chengdu
  - Research Site, Foshan
  - Research Site, Guangdong
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Jinan
  - Research Site, Langfang
  - Research Site, Nanjing
  - Research Site, Ningbo
  - Research Site, Shanghai
  - Research Site, Shijiazhuang
  - Research Site, Ürümqi
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Yantai
  - Research Site, Zhuhai

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8664R00001&attachmentIdentifier=b842b577-f113-4a2e-b502-bf4d88af6de9&fileName=D8664R00001_CSR_Synopsis.pdf&versionIdentifier=